CLINICAL TRIAL: NCT04467645
Title: The Effect of Reflexology on Sleep Quality and Fatigue in Postmenopausal Women: A Randomized Control Trial
Brief Title: The Effect of Reflexology on Sleep Quality and Fatigue in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dicle University (Other)
Responsible Party: Principal Investigator, Leyla ZENGİN AYDIN, Assistant Professor, Dicle University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: LZA2018/4
Record Dates: First submitted 2020-06-24; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Healthy; Nursing Caries
Keywords: Nurse; postmenopausal women; sleep; reflexology; fatigue
MeSH Terms: conditions — Fatigue | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: This study was conducted as a pretest-posttest trial model with a control group in order to determine the effect of reflexology applications on sleep quality and fatigue in postmenopausal women
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reflexology (Experimental): Reflexology Application: A total of twelve 30-minute reflexology sessions (2 per week)were administered to each patient.
  Interventions: Other: reflexology
- No intervention (No Intervention): No intervention was applied to the postmenopausal women in the control group.

INTERVENTIONS:
Other: reflexology — Reflexology is the stimulation of the reflex points in the hands and feet by massage, designed to provide relaxation and relief in the body.
  Arms: Reflexology

SUMMARY:
Introduction: This study was conducted to determine the effect of reflexology on sleep quality and fatigue in postmenopausal women.

DETAILED DESCRIPTION:
This study was conducted in Batıkent Family Health Center of the Ministry of Health between May-December 2018. The sample of the study consisted of 72 postmenopausal women. The data were collected by using the Introductory Information Form, Pittsburgh Sleep Quality Index and Fatigue Severity Scale. A total of 12 reflexology sessions were applied to the postmenopausal women by the researcher twice a week. No intervention was applied to the postmenopausal women in the control group.

ELIGIBILITY:
Inclusion Criteria:

* able to communicate,
* aged 50 to 65,

Exclusion Criteria:

* taking hormone replacement therapy,
* chronic diseases (such as diabetes, hypertension, and so on),
* psychiatric disease,
* diagnosed with a sleep disorder attributed to other cause
* menstruation for more than one year
* history of alcohol or drug addiction

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-09-28 (Actual)

PRIMARY OUTCOMES:
Reflexology Application, Pre-tests applied Pittsburgh Sleep Quality Index (PSQI), and Fatigue Severity Scale (FSS). | first week
  A PSQI score of 5 or higher indicates poor sleep quality. A mean total score on the FSS of four and above indicates chronic fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla ZENGİN AYDIN, Principal Investigator — Dicle University, Diyarbakır, Turkey. 21100/Diyarbakır
Locations (1):
- Leyla ZENGİN AYDIN, Diyarbakır, Sur, Turkey (Türkiye)